CLINICAL TRIAL: NCT04762758
Title: A Multi-center, Randomized, Double-blind, Placebo Controlled Phase III Study to Assess the Efficacy, Safety, and Tolerability of PXT3003 in Charcot-Marie-Tooth Type 1A (CMT1A)
Brief Title: Phase III Trial Assessing the Efficacy and Safety of PXT3003 in CMT1A Patients
Acronym: PREMIER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharnext S.C.A. (Other)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN-PXT3003-06; 2020-004805-30 (EudraCT Number)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Charcot-Marie-Tooth Disease
Keywords: Charcot Marie Tooth Type 1; Peripheral Neuropathy; PXT3003
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Peripheral Nervous System Diseases | interventions — Naltrexone; Sorbitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: PXT3003 and its matching placebo will have the same presentation, the same aspect and taste in order to be indistinguishable, and they will be supplied and used in the same conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PXT3003 (Experimental): Liquid oral solution, 10 mL twice a day, morning and evening with food
  Interventions: Drug: (RS)-baclofen, naltrexone hydrochloride and D-sorbitol
- Placebo (Placebo Comparator): Liquid oral solution, 10 mL twice a day, morning and evening with food
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: (RS)-baclofen, naltrexone hydrochloride and D-sorbitol — oral fixed dose combination
  Other Names: PXT3003
  Arms: PXT3003
Drug: Placebo — liquid oral solution
  Arms: Placebo

SUMMARY:
The study will consist of 2 periods: Double-blind Treatment and Open-Label Extension(OLE) Period.

-Double-blind Treatment Period - This will be randomized, double-blind, placebo-controlled part of the study which will be conducted in parallel groups, ie,1 group receiving the active treatment (PXT3003) and the other group receiving placebo.

Primary endpoint of the study will be assessed at Month 15.

-Open-label Extension (OLE) Period - All subjects completing Double-blind Treatment Period will be given an opportunity to enter the OLE Period of the study and receive the active treatment (PXT3003). The duration of the OLE Period will be based on Sponsor discretion, ie, Sponsor intends to keep the study open until the study drug PXT3003 is commercially available.

During this period, the long-term safety and efficacy of PXT3003 will be assessed as an exploratory objective.

Double-blind Treatment Period Objectives:

Primary:

To evaluate the efficacy of treatment with PXT3003 (a fixed-dose combination of [RS]-baclofen, naltrexone hydrochloride [HCl], and D-sorbitol) compared to placebo in subjects with Charcot-Marie-Tooth disease type 1A (CMT1A).

Secondary:

To evaluate the safety and tolerability of PXT3003 treatment in subjects with CMT1A.

Exploratory:

To characterize the relationship between plasma biomarkers and response to PXT3003 treatment.

OLE Period Objective:

Exploratory:

To evaluate the long-term safety and efficacy of PXT3003.

DETAILED DESCRIPTION:
This is an international, multi-center, randomized, double-blind, placebo-controlled, parallel-group, Phase III study of PXT3003 in subjects with CMT1A. The study will be conducted at approximately 52 sites worldwide.

This study consists of Double-blind Treatment and OLE Periods.

Double-blind Treatment Period:

Eligible subjects will be screened and randomized in a 1:1 ratio to receive either oral PXT3003 or matching placebo, 10 mL, twice daily (BID) for 15 months. In order to maximize the tolerability of (RS)-baclofen for all randomized subjects, treatment will start with a half-dose (5 mL), taken BID (morning and evening with food) during the first 2 weeks, and then will be increased to a full-dose (10 mL), taken BID (morning and evening with food) until completion of the Treatment Period at Month 15.

A total of approximately 350 subjects will be enrolled. Visits will take place at Screening (up to -35 days), Baseline (Day 1), and Months 3, 6, 9, 12, and 15. Telephone contacts will take place at weeks 2 or 3, Month 1 and Month 2, and then monthly between subsequent in-person visits. A genotyping test for the Peripheral Myelin Protein 22 (PMP22) gene duplication will take place at the Screening Visit if it is not already documented for the subject. All subjects completing the Double-blind Treatment Period of the study will be given an opportunity to enter the OLE Period at Month 15 (Visit 6). Subjects not consenting to enter the OLE Period will have their last study visit (ie, Safety Follow-up Visit, Visit 7), 30 days after their last dosing day.

The primary outcome measures modified Overall Neuropathy Limitations Score(mONLS) and the 10-Meter Walk Test (10mWT), along with the Columbia Suicide Severity Rating Scale (C-SSRS) will be evaluated at each post-randomization in-person visit. The other secondary outcome measures, exploratory outcome, and safety/tolerability assessments will be evaluated as per Schedule of Activities (SOA). A Data Safety and Monitoring Board (DSMB) will meet on a scheduled basis throughout the study to review safety data and will reconvene on an ad hoc basis as necessary.

Planned duration for sites to enroll subjects: approximately 12 months, Subject Screening Period: 35 days, Subject Treatment Period: up to 15 months, Safety Follow-up Period (for subjects not entering the OLE Period): 30 days

OLE Period:

A subject entering the OLE Period (whether the subject was randomized to oral PXT3003 or matching placebo in the Double-blind Treatment Period) will start taking a half-dose of PXT3003 (5 mL) BID (morning and evening with food) during the first 2 weeks, and then a full dose of PXT3003 (10 mL) BID (morning and evening with food) throughout the OLE Period. The visits and assessments during the OLE Period are described in the SOA.

For subjects entering the OLE Period, Screening Day will occur on the same day as Visit 6 (Month 15) of the Double-blind Treatment Period. The duration of the Treatment Period will be based on Sponsor discretion. Sponsor intends to keep the study open until the study drug PXT3003 is commercially available. Safety Follow-up Period: 30 days

ELIGIBILITY:
Double-blind Treatment Period

Inclusion Criteria:

1. Male and non-pregnant female subjects, aged 16 to 65 years with a genetically proven diagnosis of CMT1A. Notes: a) A report of a genetic test confirming PMP22 duplication and therefore a diagnosis of CMT1A must be available in the subject's record at the clinical site. b) In the absence of a report of a genetic test confirming PMP22 duplication in the subject's medical record, a confirmatory genetic test must be conducted via the central laboratory as part of Screening. c) In the exceptional case wherein subject was randomized into the study without meeting(a) or (b), an unscheduled confirmatory genetic test will be performed. In the event of a negative genetic test result, the subject will be withdrawn from the study.
2. Able to provide written informed consent/assent and comply with study procedures.
3. Mild-to-moderate severity assessed by a CMTNS-V2 score >2 and ≤18.
4. Muscle weakness in at least foot dorsiflexion on clinical assessment.
5. Ulnar nerve motor conduction time of at least 15 m/s.
6. If taking prescribed psychoactive drugs(eg, antidepressants, stimulants, tranquilizers, anti-epileptics) for CMT1A, should be on a stable dose for at least 4 weeks prior to randomization, which is not planned to be changed.
7. If taking prescribed or 'over-the-counter' analgesic medications (eg, paracetamol/acetaminophen, nonsteroidal anti-inflammatory drugs) for CMT1A, should be on a stable dose for at least 2 weeks prior to randomization, which is not planned to be changed.
8. If female, subject must be: (a) surgically sterilized via hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; or (b) of childbearing potential and using a birth control method such as:

   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Intravaginal
     * Transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Injectable
     * Implantable
   * Intrauterine device
   * Intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Sexual abstinence or (c) Of non-childbearing potential (i.e., no menses for ≥ 12 consecutive months without any other underlying medical cause)
9. If male, the subject must have had a vasectomy or must use a reliable method of birth control with their partner or total abstinence from sexual intercourse. The subject must agree to continue using their selected method of birth control with their sexual partner during the study and for 120 days after study completion.

Exclusion Criteria:

1. Subjects previously enrolled in any PXT3003 study.
2. Subjects living in the same household and enrolled in a PXT3003 study (due to potential lack of adequate storage for study material, risk of mixing treatments and potential unblinding).
3. CMT of any subtype other than 1A.
4. ONLS score of 0.
5. Known clinically significant motor or sensory abnormalities secondary to a different neurological cause (eg, diabetes, alcohol, vascular, autoimmune, neoplastic, neurodegenerative, human immunodeficiency virus, etc.). Note: subjects with diagnosis of unilateral carpal tunnel syndrome at least 1 year prior to Screening Visit, that is asymptomatic at the time of Screening Visit, will not be excluded from participating in this study.
6. Subjects who have had any surgery or have a concomitant disorder (eg, severe arthrosis) that reduces the mobility of the ankle or wrist making it, in the opinion of the investigator, difficult to assess the efficacy of the treatment. Note: subjects with surgical repair of unilateral carpel tunnel syndrome will not be excluded from participating in this study.
7. Known peripheral neuropathy, myopathy, or neuromuscular disorder of any other kind. Note: subjects with diagnosis of unilateral carpal tunnel syndrome at least 1year prior to Screening Visit, that is asymptomatic at the time of Screening Visit, will not be excluded from participating in this study.
8. Any other clinically significant and/or uncontrolled medical condition that, in the opinion of the investigator, could be a confound, may increase subject's risk, or may preclude successful participation or completion of the study.
9. Known hypersensitivity or intolerance to PXT3003( or matching placebo), including any of its active ingredients( baclofen, naltrexone, or sorbitol), and/or any of its excipients( acetate buffer, sodium methyl parahydroxybenzoate, sodium propyl parahydroxybenzoate, or isoamyl acetate).
10. Concomitant treatments including but not limited to baclofen, naltrexone, sorbitol (pharmaceutical form), opioids, potent central nervous system depressants (such as barbiturates, long-acting benzodiazepines, and neuroleptics), and potentially neurotoxic drugs such as amiodarone, chloroquine, and chemotherapeutics capable of inducing peripheral neuropathy. Subjects able to stop these medications at least 2 weeks before randomization and for the study duration may be included. Subjects with positive urine drug screen at Baseline Visit will be excluded, except for permitted use of codeine and benzodiazepines.
11. History of porphyria.
12. Diagnosis or history of substance use disorder by Diagnostic and Statistical Manual of Mental Disorders-5th Edition criteria within the past 12 months.
13. Medical or recreational use of marijuana in the 3 months prior to the Screening Visit.
14. Active suicidality (eg, any suicide attempts within the past 12 months or any current suicidal intent, including a plan, as assessed by the C SSRS score of "YES" on questions 4 or 5; and/or based on clinical evaluation by the investigator).
15. Currently active major depression, as determined by a Beck Depression Inventory-II (BDI-II) score ≥20.
16. Currently lactating, pregnant, or planning on becoming pregnant during the study.
17. Alanine aminotransferase or aspartate aminotransferase levels greater than 2 times the upper limit of normal.
18. Significant renal impairment as determined by glomerular filtration rate of less than 50 mL/min.
19. Subject has participated in an investigational drug or device study within 30 days prior to the Screening Visit or plans to participate in an investigational drug or device study during the course of this study.
20. Subject is a dependent and/or relative of the Sponsor or Principal Investigator.

OLE Period

Inclusion Criteria:

1. Able to provide written informed consent/assent and comply with study procedures.
2. If female, subject must be (a) surgically sterilized via hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; or (b) of childbearing potential and using a birth control method such as:

   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Intravaginal
     * Transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Injectable
     * Implantable
   * IUD
   * IUS
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Sexual abstinence or (c) of non-childbearing potential (ie, no menses for ≥12 consecutive months without any other underlying medical cause).
3. If male, the subject must have had a vasectomy or must use a reliable method of birth control with their partner or total abstinence from sexual intercourse. The subject must agree to continue using their selected method of birth control with their sexual partner during the study and for 120 days after study completion.

Exclusion Criteria:

1. Any clinically significant and/or uncontrolled medical condition that, in the opinion of the investigator, could be a confound factor, may increase subject's risk, or may preclude successful participation or completion of the study.
2. Concomitant treatments including but not limited to baclofen, naltrexone, sorbitol (pharmaceutical form) other than PXT3003 taken in the Double-blind Treatment Period of this study, opioids, potent CNS depressants (such as barbiturates, long-acting benzodiazepines, and neuroleptics), and potentially neurotoxic drugs such as amiodarone, chloroquine, and chemotherapeutics capable of inducing peripheral neuropathy. Subjects able to stop these medications at least 2 weeks before randomization and for the study duration may be included.
3. Diagnosis or history of substance use disorder by Diagnostic and Statistical Manual of Mental Disorders-5ᵗʰ Edition criteria within the past 12 months.
4. Active suicidality (eg, any suicide attempts within the past 12 months or any current suicidal intent, including a plan, as assessed by the C-SSRS score of "YES" on questions 4 or 5; and/or based on clinical evaluation by the investigator).
5. Currently active major depression, as determined by a BDI-II score ≥20.
6. Currently lactating, pregnant, or planning on becoming pregnant during the study.
7. ALT or AST levels greater than 2 × ULN relative to Baseline.
8. Estimated GFR of less than 50 mL/min.

Note: PXT3003 will be dispensed to all subjects before laboratory results are available, and if the laboratory results are out of range, ie, subject meeting the exclusion criteria, the subject will be called immediately to stop taking PXT3003. One retest within 4 weeks may be performed in consultation with the Medical Monitor if any of the above laboratory abnormalities are found. In case of eligibility determination after the retest, subjects will restart taking 2 weeks of half dose of PXT3003.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-04-19 (Estimated); Study Completion 2024-04-19 (Estimated)

PRIMARY OUTCOMES:
modified Overall Neuropathy Limitation Scale (mONLS) | From Baseline to Month 15
  The modified ONLS is a disability scale that was derived and improved from the Overall Disability Sum Score to measure limitations in the everyday activities of the upper limbs (rated on 5 points) and the lower limbs (rated on 7 points).38 The total score goes from 0 (no disability) to 12 (maximum disability). Lower values in the ONLS indicate a better clinical condition.

SECONDARY OUTCOMES:
10-Meter Walk Test | From Baseline to Month 15
  The 10mWT is simple to administer, standardized, and valid performance evaluation of functional mobility and gait that has been proven reliable in neurologic disorders, including CMT. Results recorded are the time to walk 10 meters and the number of steps performed.
Quantified Muscular Testing (QMT) (bilateral foot dorsiflexion dynamometry) | From Baseline to Month 15
  QMT is used to evaluate motor strength in CMT1A.The following muscles will be evaluated: tibialis anterior (right and left). The best value on three consecutive and reproducible tests will be collected in the electronic Case Record Form (eCRF) for each muscle.
Patient Global Impression of Severity (PGI-S) | From Baseline to Month 15
  The PGI-S is a validated tool that is used to rate the severity of a specific condition. Subjects will rate their health status over the past week. The PGI-S is a 1-item questionnaire on a 5-point scale and subjects will be asked to rate the severity of their condition from "None" (Score = 1) to "Very Severe" (Score = 5). Assessments obtained over the course of the study will be compared to baseline, prior to initiation of treatment.
Patient Global Impression of Change (PGI-C) | From Baseline to Month 15
  The PGI-C scale is a validated generic tool for assessment of overall change in the severity of illness following treatment. Subjects will rate how they feel now compared with how they felt before receiving study drug on a 7-point scale where 1 is "Very much improved" and 7 is "Very much worse".
CMTNS-V2 | From Baseline to Month 15
  CMTNS is a specific scale designed to assess severity of impairment in CMT disease. Although not completely validated, it provides a single and reliable measure of CMT severity. It is a 36-point scale based on 9 items: 5 of them quantify impairment (sensory symptoms, pin sensibility, vibration, arm, and leg strength), 2 activity limitations (motor symptoms arms and legs) and 2 electrophysiological data (amplitudes of ulnar compound muscle action potential and sensory nerve action potential). Increased scores indicate a worsening of the function: the scores categorize a disability as mild (0 to10), moderate (11 to 20) and severe (21 to 36).
  A modified version 2 (CMTNS-V2) was issued in 2011 to attempt to reduce floor and ceiling effects and to standardize patient assessment.
QMT (hand grip) | From Baseline to Month 15
  QMT is used to evaluate motor strength in CMT1A. The following muscles will be evaluated: hand grip (right and left). The best value on three consecutive and reproducible tests will be collected in the eCRF for each muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Sharam Attarian, MD, Principal Investigator — CHU la Timone, Marseille , France; Mario Saporta, MD, Principal Investigator — University of Miami Miller School of Medicine, USA
Locations (50):
- United States (20):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Department of Psychiatry and Biobehavioral Sciences, Los Angeles, California
  - UC Davis Health Department of Physical Medicine and Rehabilitation, Sacramento, California
  - Hospital for Special Care, New Britain, Connecticut
  - University of Florida Clinical Research Center, Gainesville, Florida
  - University of Miami Leonard M. Miller School of Medicine, Miami, Florida
  - Advent Health Medical Group Neurology Orlando, Orlando, Florida
  - University of Kansas Medical Center Research Institute, Fairway, Kansas
  - Massachusetts General Hospital Neuromuscular Diagnostic Center, Boston, Massachusetts
  - University of Minnesota Health, Minneapolis, Minnesota
  - MU Health Care Neurology and Sleep Disorders Clinic, Columbia, Missouri
  - Hackensack Meridian Health Hackensack University Medical Center, Hackensack, New Jersey
  - Colombia University Department of Neurology, New York, New York
  - UNC Department of Neurology Peripheral Neuropathy Center, Chapel Hill, North Carolina
  - Atrium Health Neurosciences Institute, Charlotte, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Neurology, Springfield, Oregon
  - National Neuromuscular Research Institute, Austin, Texas
  - Neurology Clinic at University of Washington Medical Center, Seattle, Washington
  - Providence St. Luke's Rehabilitation Medical Center, Spokane, Washington
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Canada (5):
  - Ottawa Hospital Research Institute- Neuromuscular Research Centre, Ottawa, Ontario
  - UHN Toronto General Hospital Krembil Neuroscience Centre, Toronto, Ontario
  - CIUSS de Saguenay-Lac-Saint-Jean Centre d'etudes Cliniques, Chicoutimi, Quebec
  - Montreal Neurological Institute and Hospital-Clinical Research Unit, Montreal, Quebec
  - CHU de Quebec-Universite Laval- Hopital Enfant-Jesus, Québec, Quebec
- Rigshospitalet, University of Copenhagen Copenhagen Neuromuscular Center, Copenhagen, Denmark
- France (6):
  - Centre de Reference des Maladies Neuromusculaires AOC Service de Neurologie, CHU d'Angers, Angers
  - Centre de reference des maladies neuromusculaires AOC Hopital Pellegrin CHU de Bordeaux, Bordeaux
  - CHU de Lille Hôpital Salengro, Lille
  - Service de Neurologie et Maladies Neuromusculaires, CHU de Marseille - Hopital La Timone, Marseille
  - Association lnstitut de Myologie Hopital Pitie-Salpetriere Service de Neuro-Myologie, Paris
  - Centre d'investigation Clinique CHU de Strasbourg Hopital de Hautepierre, Strasbourg
- Germany (5):
  - University Hospital RWTH Aachen, Department of Neurology and Institute for Neuropathology, Aachen
  - University Medical Centre Goettingen, Dept. of Clinical Neurology, Göttingen
  - Friedrich-Baur-Institut, Neurologische Klinik und Poliklinik Ludwig-Maximilians-Universität, München
  - University Hospital Muenster UKM Department of Neurology, Münster
  - Universitätsklinikum Tübingen Crona Kliniken Neuromuskuläres Zentrum, Tübingen
- Israel (3):
  - Hadassah Ein Kerem University Medical Center Department of Neurology, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Universitaria San Martino Universita Degli Studi di Genova Clinica Neurologica, Genova
  - Azienda Ospedaliera Universitaria Policlinico "G. Martino" di Messina, Messina
  - University of Naples Federico II, Naples
  - Tor Vergata University of Rome, Rome
  - University Hospital GB Rossi UOC Neurologia B, AOUI Verona Department of Neuroscience, Biomedicine and Movement Sciences, Verona
- Spain (4):
  - Hospital Universitario Clinico San Carlos, Madrid
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fé, Valencia

IPD SHARING:
Plan to Share IPD: No